CLINICAL TRIAL: NCT02537340
Title: The Use of PET/MR for Initial Staging of Rectal Cancer Patients With Extramural Vascular Invasion Detected by MR (EMVI-MR)
Brief Title: PET/MR for Staging Rectal Cancer Patients With and Without EMVI-MR
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Marcelo Araujo Queiroz, MD, Instituto do Cancer do Estado de São Paulo
Other Study IDs: NP796/15
Record Dates: First submitted 2015-08-30; First posted 2015-09-01 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Rectal Neoplasms
Keywords: PET/MR; MRI; Rectal cancer; EMVI; FDG
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- EMVI-MR positive: Patients with primary rectal cancer and extramural vascular invasion detected by staging MR
- EMVI-MR negative: Patients with primary rectal cancer and without extramural vascular invasion detected by staging MR

SUMMARY:
The hypothesis to be proven with this study is that the use of PET/MR on the initial staging of rectal cancers in patients with extramural vascular invasion detected by MR will detect more lesions than conventional work-up and will significantly impact on therapeutic decision, improving disease free and overall survival.

DETAILED DESCRIPTION:
The accurate staging of rectal cancer is essential to define therapy and for prognosis assessment. Imaging modalities usually provide useful information for pre-operative planning of primary tumour resection and may indicate the need of neoadjuvant treatment. It is recommended the use of magnetic resonance imaging (MRI) for local staging and computed tomography (CT) of chest, abdomen and pelvis for detection of distant metastasis. Patients with rectal cancer and vascular invasion might benefit from an intensive pre-operative staging in order to early detect distant metastasis, favouring a better therapeutic planning. There is no consensus regarding the use of PET/MR for initial staging of patients with rectal cancer. It has been shown that although changing pattern's in patients' stage, the use of PET/MR for colorectal cancers did not impact disease management. New studies are required for identifying the subgroup of patients with changes in the pre-operative MR that might benefit from the use of PET/MR for initial staging of rectal cancers.

Patients with rectal cancer will undergo pelvic MR, whole-body CT and whole-body PET/MR. According to the tumour characteristics on MR, there will be defined two group of patients: with EMVI-RM (group A) and without EMVI-MR (group B). The whole-body CT and PET/MR will be evaluated for the detection of loco-regional lymph nodes disease and distant metastasis. The total number of lesions and their respective sites will be recorded and compared for each method. The PET/MR management impact will be determined from the medical record or by direct contact with the treating clinician. The impact of PET/MR on management will be defined as high (the treatment modality or intent was changed), medium (the treatment modality or intent remained unchanged, although the method of treatment delivery or planned diagnostic procedure was changed), low (PET/MR results were consistent with planned management, and treatment modality or intent was unchanged), or none (the management plan was not changed, despite being inconsistent with the PET/MR stage-that is, PET/MR results were ignored). Overall survival will be used to evaluate prognostic significance. Clinical follow-up will be performed 3 monthly for 2 years. Imaging and, eventually biopsy, will be performed to evaluate symptoms or signs suggestive of residual or recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* No contraindication to MRI (eletromagnetic devices, claustrophobia);
* No contraindication to PET/MR (hyperglycemia, claustrophobia);
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Local resection of rectal tumor;
* Non-colorectal synchronic lesion;
* Previous treatment (chemo or radiation therapy) for rectal cancer;
* Renal insufficiency;
* Pregnancy, lactation or inadequate contraception
* Known allergy to contrast media (CT, MR or PET);
* Blood glucose level higher than 150 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven rectal cancer.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Detection rate | 12 months
  Number of metastatic lesions detected

SECONDARY OUTCOMES:
Clinical Impact | 12 months
  Measured by change in patient's therapy through questionnaire applied to referring physician
Progression-free survival | 36 months
  Measured in terms of loco-regional or distant recurrence by 3 years.
Overall survival | 36 months
  Measured in terms of death related to disease by 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Buchpiguel, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Queiroz MA, Ortega CD, Ferreira FR, Capareli FC, Nahas SC, Cerri GG, Buchpiguel CA. Value of Primary Rectal Tumor PET/MRI in the Prediction of Synchronic Metastatic Disease. Mol Imaging Biol. 2022 Jun;24(3):453-463. doi: 10.1007/s11307-021-01674-1. Epub 2021 Nov 9. PMID 34755248
- [Derived] Queiroz MA, Ortega CD, Ferreira FR, Nahas SC, Cerri GG, Buchpiguel CA. Diagnostic accuracy of FDG-PET/MRI versus pelvic MRI and thoracic and abdominal CT for detecting synchronous distant metastases in rectal cancer patients. Eur J Nucl Med Mol Imaging. 2021 Jan;48(1):186-195. doi: 10.1007/s00259-020-04911-x. Epub 2020 Jun 20. PMID 32561971